CLINICAL TRIAL: NCT04212026
Title: Irreversible Electroporation (IRE) Followed by Nivolumab in Patients With Metastatic Pancreatic Cancer: a Multicenter Single-arm Phase II Trial
Brief Title: Irreversible Electroporation (IRE) Followed by Nivolumab in Patients With Metastatic Pancreatic Cancer.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficult recruitement
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: St. Clara Research Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDAC-IRE
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: metastatic Pancreatic Cancer; Irreversible electroporation (IRE); nivolumab; Phase II trial
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a pilot, multicenter, single-arm phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab treatment will be given every 2 weeks at a standard flat dose of 240 mg for a total of 5 doses, and the IRE procedure will be performed using the standard setting to ablate tumors at the level of the liver that is well tolerated by the patients. Two weeks after the last dose of nivolumab ("Week 8"), radiological restaging will be performed (="Week 10").
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — The patients start treatment with nivolumab on day 1 after IRE and will be given nivolumab at a flat dose of 240 mg every 2 weeks (q2wk) for 5 cycles until Week 8.

SUMMARY:
This proof of concept trial aims to assess whether the combination of IRE with Nivolumab is safe and effective to treat metastatic pancreatic cancer, based on the available preliminary evidence that IRE is able to cause a systemic anti-tumor immune response (i.e. abscopal effect), which may enhance the effect of subsequent Nivolumab treatment. In addition, the trial aims to clarify the systemic effects of IRE over time and thereby to provide more insight in the mechanism of work of the technique.

DETAILED DESCRIPTION:
The prognosis of patients newly diagnosed with pancreatic ductal adenocarcinoma (PDAC) is extremely poor with a 5-year overall survival rate of less than 5%. To improve this dismal outcome, new treatment approaches are urgently needed. So far, immune-checkpoint therapy was not successful in patients with PDAC. Given the poor response to conventional chemotherapy, there is an imperative need to make PDACs amenable to immune-checkpoint therapy. Irreversible electroporation (IRE) is a relatively novel and safe ablation technique that destroys tumors by using apoptosis-inducing electrical currents inducing local and systemic pro-inflammatory cytokine expression and enhances the presence of cytotoxic CD8+ T-cells, while the apoptotic cell material preserves neo-antigen properties detectable by dendritic cells. This effect might be further enhanced by immune-checkpoint therapy.

The rationale of our study is to convert immunologically cold PDACs into hot PDACs by triggering an enhanced local and systemic immune response. We hypothesize that among patients with metastatic PDAC, the IRE of one liver metastasis followed by the administration of an immune-checkpoint inhibitor leads to a measurable radiological response in a selected non-treated liver metastasis. Furthermore, we hypothesize that the immune response is both local in the form of tumor infiltrating lymphocytes (TILS) and an immunologically activated tumor microenvironment in the IRE-treated metastasis, as well as systemic as evidenced by an abscopal response in the IRE-untreated metastatic and primary site.

The objective of the trial is to examine whether for patients with metastatic PDAC the combination of IRE of one liver metastasis followed by the administration of five doses of nivolumab leads to a measurable radiological response in a selected non-treated liver metastasis.

To demonstrate that the trial treatment leads to a measurable immune response, multiple translational research projects will assess the effect of IRE and nivolumab on the development of the local and peripheral tumor immune response over time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH GCP E6(R2) regulations before registration and prior to any trial specific procedures.
* Pathologically proven PDAC with liver metastases either by histology or cytology.
* Liver metastases fulfilling the following criteria:

  1. measurable per RECIST v 1.1 (Appendix 1), AND
  2. at least two metastases ≥ 1 cm AND
  3. percutaneously accessible for repeat biopsy, AND
  4. one of the biopsied metastases can be treated with IRE.
* At least stable disease after the completion of 10-24 weeks of first line standard chemotherapy (either (m)FOLFIRINOX or Gemcitabine/Abraxane) as confirmed by tumor assessment within 21 days prior to registration OR at least stable disease after the completion of 10-24 weeks of second line standard chemotherapy (either (m)FOLFIRINOX or Gemcitabine/Abraxane) as confirmed by tumor assessment within 21 days prior to registration. The choice of chemotherapy regimen is based on the decision of the treating medical oncologist.
* Patients with a prior malignancy and treated with curative intention are eligible if all treatment of that malignancy was completed at least 2 years before registration and the patient has no evidence of that disease at registration. Note: Less than 2 years is acceptable for malignancies with low risk of recurrence and/or no late recurrence.
* Patients must be willing to participate in the translational research part of the trial and to undergo a tumor biopsy of the primary tumor and of the two metastatic sites in the liver before trial treatment and after five cycles of nivolumab treatment.
* Patients must be willing to travel to the hospital where IRE and biopsy will be performed (Claraspital Basel).
* Age ≥ 18 years
* WHO performance status 0-1
* Life expectancy ≥4 months
* Adequate bone marrow function: neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 80 g/L
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST and ALT ≤ 3 x ULN.
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2 (according to CKD-EPI formula).
* Adequate coagulation function: INR ≤ 1.5 x ULN (the ULN for INR is defined with the value 1.2 for all sites, in case no ULN is documented in the lab certificates/sheets). In case patient is under anti-vitamin K treatment, INR >1.5 x ULN is allowed; however, the patient has to be switched to LMWH treatment prior to any trial intervention.
* Women of childbearing potential must use effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 5 months after the last dose of nivolumab. A negative pregnancy test before inclusion into the trial is required for all women of childbearing potential (for nivolumab product information).
* Men agree not to donate sperm or to father a child during trial treatment and until 7 months after the last dose of nivolumab (for nivolumab product information).

Exclusion criteria:

* Clinically significant ascites that is not controllable.
* Prior radiotherapy to any PDAC disease site.
* Prior treatment with any immune checkpoint inhibitor.
* Concomitant or recent (within 100 days of registration) treatment with any other experimental drug (enrollment in another clinical trial).
* Concomitant use of other anti-cancer drugs or radiotherapy.
* Severe or uncontrolled concurrent illness, such as cardiovascular disease (congestive heart failure NYHA III or IV; unstable angina pectoris, history of myocardial infarction within the last six months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension.
* Known history of human immunodeficiency virus (HIV) or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (i.v.) antimicrobial treatment.
* Known history of tuberculosis, known history of primary immunodeficiency, known history of allogeneic organ transplant, receipt of live attenuated vaccine within 30 days prior to registration.
* Concomitant or prior use of immunosuppressive medication within 30 days of registration, with the exceptions of intranasal and inhaled corticosteroids, or systemic corticosteroids which must not exceed 10 mg/day of prednisone (or a dose equivalent corticosteroid), and the premedication for chemotherapy
* Concomitant need for full anticoagulation treatment that cannot be stopped or bridged for the performance of the biopsy/IRE procedures Note: Aspirin or other acetylsalicylic acid containing drugs (up to 300 mg/day) are allowed
* Any concomitant drugs contraindicated for use with the trial treatment according to the approved product information
* Known hypersensitivity to nivolumab or to any component of nivolumab, to stainless steel or to contrast agents.
* Any other serious underlying medical (in particular coagulation deficiencies), psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) after the 5th dose of nivolumab of the reference liver metastasis that was not biopsied. | At 2-4 weeks after the 5th dose of nivolumab
  The objective response rate (ORR) according to RECIST v1.1 after the 5th dose of nivolumab of the reference liver metastasis that was not biopsied, assessed 2-4 weeks after the 5th dose of nivolumab, defined as proportion of patients achieving Complete Response (CR) or Partial Response (PR). The assessment will be based on re-staging the patients with a CT-scan 2-4 weeks after the 5th dose of nivolumab. Patients without tumor assessment 2-4 weeks after the 5th dose of nivolumab will be counted as non-responders.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) after the 5th dose of nivolumab of the primary tumor site (pancreas). | At 2-4 weeks after the 5th dose of nivolumab
  The ORR according to RECIST v1.1 after the 5th dose of nivolumab of the primary tumor site (pancreas), assessed 2-4 weeks after the 5th dose of nivolumab, defined as percentage of patients achieving Complete Response (CR) or Partial Response (PR). Patients without tumor assessment 2-4 weeks after the 5th dose of nivolumab will be counted as non-responders.
ORR after the 5th dose of nivolumab of the IRE-treated liver metastasis | At 2-4 weeks after the 5th dose of nivolumab
  The ORR according to RECIST v1.1 after the 5th dose of nivolumab of IRE-treated liver metastasis, assessed 2-4 weeks after the 5th dose of nivolumab, defined as percentage of patients achieving CR or PR. Patients without tumor assessment 2-4 weeks after the 5th dose of nivolumab will be counted as non-responders.
ORR based on best overall response | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  The ORR based on best overall response according to RECIST v1.1, assessed at any time between registration and disease progression by RECIST v1.1, death, or subsequent anticancer therapy, whichever occurs first, defined as percentage of patients achieving CR or PR.
Immune ORR (iORR) based on best overall immune response | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  The immune ORR (iORR) based on best overall immune response according to iRECIST, assessed at any time between registration and disease progression by iRECIST, death, or subsequent anticancer therapy, whichever occurs first, defined as percentage of patients achieving CR, PR, iCR or iPR.
Progression free survival (PFS) | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  Progression-free survival (PFS), defined as the time from registration until progression according to RECIST v1.1 or death from any cause, whichever occurs first.
Immune PFS (iPFS) | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 4 years after registration
  Immune PFS (iPFS), defined as the time from registration until progression according to iRECIST (first iUPD without documented iSD, iPR or iCR thereafter) or death from any cause, whichever occurs first.
  Patients without event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of the last tumor assessment showing non-progression (before the start of the new therapy, if any).
Overall survival (OS) | From the date of registration until the date of death, assessed up to 4 years after registration
  Overall survival (OS), defined as time form registration to death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known alive.
Adverse events | From the date of registration to 100 days after last trial treatment
  Adverse events, assessed according to NCI CTCAE v5.0 and Clavien-Dindo Classification for procedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Worni, MD, Study Chair — Clarunis - St. Clara Hospital and University Hospital Basel
Locations (3):
- Switzerland (3):
  - Lindenhofspital, Bern, Canton of Bern
  - St. Claraspital, Basel
  - UniversitätsSpital Zürich, Zurich